CLINICAL TRIAL: NCT06657456
Title: Nutritional Intervention Study of the Effect of a Phytosterol-rich Extract on Lipid Profile.
Brief Title: Impact of Phytosterol-Rich Extract on Lipid Profile
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Desirée Victoria Montesinos (Other)
Collaborators: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Sponsor-Investigator, Desirée Victoria Montesinos, Principal Investigator, Universidad Católica San Antonio de Murcia
Organization: Universidad Católica San Antonio de Murcia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CE102401
Record Dates: First submitted 2024-10-19; First posted 2024-10-24 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Cholesterol, Elevated; Hypercholesterolaemia; Lipid Metabolism Disorders; Dyslipidemias
Keywords: Cholesterol; Cholesterol, Elevated; Hypercholesterolaemia; Lipid Metabolism Disorders; Dyslipidemias
MeSH Terms: conditions — Hypercholesterolemia; Lipid Metabolism Disorders; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Consumption of dietary supplement capsules for 56 days.
  Interventions: Dietary Supplement: Phytosterol-rich extract
- Control Group (Placebo Comparator): Identically appearing placebo capsules consumed for 56 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Phytosterol-rich extract — Experimental product: extract rich in phytosterols
  Arms: Experimental
Dietary Supplement: Placebo — Product with identical characteristics to the experimental product.
  Arms: Control Group

SUMMARY:
The aim of this randomized, parallel, two-arm, placebo-controlled, triple-blind clinical trial is to evaluate the efficacy of a phytosterol- and phytostanol-rich extract on lipid profile parameters in individuals with hypercholesterolemia, focusing primarily on total cholesterol and LDL cholesterol levels.

DETAILED DESCRIPTION:
The duration of the study will be 56 days during which the investigational product or placebo will be consumed according to the assignment.

Subjects will be randomized to each of the study arms (consumption of the experimental product or control product).

ELIGIBILITY:
Inclusion Criteria:

* Adults (age > 18 YO)
* Total cholesterol levels at screening ≥ 200 mg/dL

Exclusion Criteria:

* History of allergic hypersensitivity or poor tolerance to any component of the products under study.
* Use of prescribed medication which may interfere with study measurements.
* Unwillingness or inability to comply with clinical trial procedures.
* Subjects whose condition makes them ineligible for the study at the investigator's discretion.
* Pregnant or having the wish to become pregnant, or lactating.
* Recent participation in another nutritional or medical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Blood lipid profile | Day 1, at 28 and 56 days
  Includes total cholesterol, LDL-cholesterol, HDL-cholesterol and triglycerides

SECONDARY OUTCOMES:
Anthropometric parameters | Day 1, at 28 and 56 days
  Body weight (Kg), body mass index (kg/m^2) and waist circumference (cm)
Body composition measures | Day 1, at 28 and 56 days
  Fat-free mass (Kg) and fat mass (Kg)
Oxidation markers | Day 1, at 28 and 56 days
  Measurement of oxidized LDL
Dietary Intake | Day 1, at 28 and 56 days
  Registration and subsequent nutritional evaluation with 3-day food frequency questionnaire (FFQ).
Adherence to the Mediterranean diet | Day 1, at 28, and 56 days
  Measurement of adherence to the Mediterranean diet by the MEDAS questionnaire.
Blood pressure | Day 1, at 28 and 56 days
  Systolic blood pressure and diastolic blood pressure (mmHg).
Physical Activity | Day 1, at 28 and 56 days
  Measured by IPAQ/GPAQ questionnaire.
Liver safety variables | Day 1, at 28 and 56 days
  It is a blood test that measures liver enzymes, such as GPT (ALT) and GOT (AST), to evaluate liver function.

CONTACTS AND LOCATIONS:
Overall Officials: Desirée Victoria Montesinos, Principal Investigator — Universidad Católica San Antonio de Murcia; Ana Mª García Muñoz, Principal Investigator — Universidad Católica San Antonio de Murcia
Locations (1):
- UCAM San Antonio Catholic University of Murcia, Murcia, Murcia, Spain